CLINICAL TRIAL: NCT01287988
Title: Follow-up Study to Assess Visual Function in Subset of Patients Who Have Previously Participated in the TG-MV-006 and TG-MV-007 Ocriplasmin Studies.
Status: Completed | Type: Observational
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Other Study IDs: TG-MV-012
Record Dates: First submitted 2011-01-24; First posted 2011-02-02 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2014-04

CONDITIONS: Symptomatic Vitreomacular Adhesion
MeSH Terms: interventions — microplasmin

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ocriplasmin: Subjects who were exposed to a single intravitreal injection of 125µg of ocriplasmin in a previous phase III study (TG-MV-006 or TG-MV-007)
  Interventions: Drug: ocriplasmin
- Placebo: Subjects who were exposed to a single intravitreal injection of placebo in a previous phase III study (TG-MV-006 or TG-MV-007)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ocriplasmin — Subjects were exposed to a single intravitreal injection of 125µg of ocriplasmin in a previous phase III study TG-MV-006 or TG-MV-007
  Groups: Ocriplasmin
Drug: placebo — Subjects were exposed to a single intravitreal injection of placebo in a previous phase III study TG-MV-006 or TG-MV-007
  Groups: Placebo

SUMMARY:
The primary objective of this study is to assess visual function in up to 44 patients who have previously participated in either of the placebo controlled, ocriplasmin Phase III studies (TG-MV-006 or TG-MV-007).

DETAILED DESCRIPTION:
Non-interventional follow up study consisting of 1 patient visit to perform assessments to assess long term visual function

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient prior to inclusion in the follow-up study
* Previous participation in either of the placebo controlled, ocriplasmin Phase III studies (TG-MV-006 or TG-MV-007)

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have previously participated in either of the ocriplasmin Phase III studies (TG-MV-006 or TG-MV-007)
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Evidence of clinically significant abnormality in visual function, including Best Corrected Visual Acuity (BCVA), Spectral Domain Optical Coherence Tomography (SD-OCT) abnormality, and/or Electroretinography (ERG) abnormality | Visit 1
  Consenting patients will attend one visit, at which an ocular history, visual acuity (ETDRS) and full ophthalmologic assessment, as well as SD-OCT, and ERG assessment will be obtained. All SD-OCTs and ERGs will be centrally read by a masked and independent central reader.

CONTACTS AND LOCATIONS:
Locations (2):
- Retinal Consultants of Houston, Houston, Texas, United States
- Universitaire Ziekenhuizen K.U. Leuven, Leuven, Belgium